CLINICAL TRIAL: NCT00608491
Title: CARdiorenal REScue Study in Acute Decompensated Heart Failure: CARRESS
Brief Title: Effectiveness of Ultrafiltration in Treating People With Acute Decompensated Heart Failure and Cardiorenal Syndrome (The CARRESS Study)
Acronym: CARRESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Nuwellis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00018064; U01HL084904-04 (NIH); U01HL084904 (NIH); 522
Record Dates: First submitted 2008-01-25; First posted 2008-02-06 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-05

CONDITIONS: Heart Failure
Keywords: Acute Decompensated Heart Failure; Acute Decompensated Heart Failure With Cardiorenal Syndrome; Cardiorenal Syndrome; Persistent Congestion; Ultra Filtration
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome | interventions — Ultrafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stepped pharmacologic care (Active Comparator): Stepped care will provide treating physicians with guidelines for the intensification of diuretic therapy and the possible use of vasodilators and inotropes.
  Interventions: Drug: Stepped pharmacologic care
- Ultrafiltration (Experimental): All loop diuretics will be discontinued. Treatment will involve slow continuous ultrafiltration until an optimal volume status has been achieved. Ultrafiltration therapy will be initiated after the placement of appropriate intravenous access and will continue until the participant's signs and symptoms of congestion have been optimized. Fluid status will be managed exclusively by ultrafiltration using the Aquadex system 100 (CHF Solutions, Inc.) according to the manufacturer's specifications. The use of vasodilators or inotropic agents will be prohibited unless deemed necessary for rescue therapy.
  Interventions: Device: Ultrafiltration

INTERVENTIONS:
Drug: Stepped pharmacologic care — Stepped care will provide treating physicians with guidelines for the intensification of diuretic therapy and the possible use of vasodilators and inotropes.
  Arms: Stepped pharmacologic care
Device: Ultrafiltration — All loop diuretics will be discontinued. Treatment will involve slow continuous ultrafiltration until an optimal volume status has been achieved. Ultrafiltration therapy will be initiated after the placement of appropriate intravenous access and will continue until the participant's signs and symptoms of congestion have been optimized. Fluid status will be managed exclusively by ultrafiltration using the Aquadex system 100 (CHF Solutions, Inc.) according to the manufacturer's specifications. The use of vasodilators or inotropic agents will be prohibited unless deemed necessary for rescue therapy.
  Arms: Ultrafiltration

SUMMARY:
Heart failure is a serious condition in which the heart's ability to pump blood through the body is impaired, often making a person feel weak or fatigued. When a person's condition worsens to the point of hospitalization, that person is said to have acute decompensated heart failure (ADHF). Abnormal kidney function in association with cardiac distress, known as cardiorenal syndrome, is a common complication of heart failure and causes further medical problems and need for hospitalization. While there are various effective treatments for heart failure, more research is needed to determine the best treatment for targeting both ADHF and cardiorenal syndrome. This study will compare the safety and effectiveness of ultrafiltration versus standard medical drug therapy in improving renal function and relieving fluid buildup in people hospitalized with ADHF and cardiorenal syndrome.

DETAILED DESCRIPTION:
Heart failure is a common condition that affects approximately 5 million people in the United States, with 550,000 new cases diagnosed each year. Common symptoms of heart failure include swelling and fluid buildup in the legs, feet, and/or lungs; shortness of breath; coughing; elevated heart rate; change in appetite; and fatigue. If left untreated, the condition of the heart may deteriorate so far that the person undergoes ADHF. The number of hospitalizations attributed to ADHF has risen significantly, with many people readmitted soon after discharge because of recurring symptoms or further medical complications, such as cardiorenal syndrome. Current heart failure treatments focus on removing excess fluid buildup, often by increasing urination with diuretic medications or by draining directly from the veins. Direct drainage from the veins, also known as ultrafiltration, may be the more effective method for treating people with ADHF and cardiorenal syndrome. This study will compare the safety and effectiveness of ultrafiltration versus standard medical drug therapy in improving renal function and relieving fluid buildup in people hospitalized with ADHF and cardiorenal syndrome.

Participation in this study will last 60 days. All potential participants will undergo initial screening, which will include a medical history, physical exam, blood draws, measurements of fluid intake and urine output, and questionnaires. These same evaluations and procedures will be repeated at various points during the hospital stay. Eligible participants will be randomly assigned to receive standard medical drug therapy or fluid removal by ultrafiltration. Standard medical drug therapy will involve the intravenous delivery of diuretics and possibly other doctor-recommended medications. Ultrafiltration will involve intravenously removing blood, passing it through an ultrafiltration device, and then returning the blood to the participant. During ultrafiltration, participants will be treated with a blood thinner through the IV, as well.

Follow-up assessments will occur at Days 30 and 60 after treatment. Follow-up assessments will include measurements of fluid intake, urine output, and vital signs; blood draws; physical exams; and questions about medications and status of recovery.

ELIGIBILITY:
Inclusion criteria:

* age 18 or older
* admitted to the hospital with a primary diagnosis of decompensated heart failure
* onset of cardiorenal syndrome after hospitalization or pre-hospitalization
* after hospitalization - onset of cardiorenal syndrome after hospitalization must occur within 10 days from the time of admission after receiving IV diuretics
* pre-hospitalization - onset of cardiorenal syndrome pre-hospitalization must occur within 12 weeks of the index hospitalization in the setting of escalating doses of outpatient diuretics
* persistent volume overload

Exclusion criteria:

* intravascular volume depletion based on investigator"s clinical assessment
* acute coronary syndrome within 4 weeks
* indication for hemodialysis
* creatinine > 3.5 mg per deciliter at admission to the hospital
* systolic blood pressure < 90 mmHg at the time of enrollment
* alternative explanation for worsening renal function such as obstructive nephropathy,contrast induced nephropathy, acute tubular necrosis
* Hematocrit > 45%
* poor venous access
* clinical instability likely to require the addition of intravenous vasoactive drugs including vasodilators and/or inotropic agents
* allergy or contraindications to the use of heparin
* the use of iodinated radio contrast material in the last 72 hours or anticipated use of IV contrast during the current hospitalization
* known bilateral renal artery stenosis
* active myocarditis
* hypertrophic obstructive cardiomyopathy
* severe valvular stenosis
* complex congenital heart disease
* sepsis or ongoing systemic infection
* enrollment in another clinical trial involving medical or device based interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2008-03; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry L. Lee, PhD, Principal Investigator — Duke Clinical Research Institute
Locations (9):
- United States (8):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Morehouse School of Medicine, Atlanta, Georgia
  - Minnesota Heart Failure Network, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Health Sciences Center, Murray, Utah
  - University of Vermont - Fletcher Allen Health Care, Burlington, Vermont
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Result] Bart BA, Goldsmith SR, Lee KL, Givertz MM, O'Connor CM, Bull DA, Redfield MM, Deswal A, Rouleau JL, LeWinter MM, Ofili EO, Stevenson LW, Semigran MJ, Felker GM, Chen HH, Hernandez AF, Anstrom KJ, McNulty SE, Velazquez EJ, Ibarra JC, Mascette AM, Braunwald E; Heart Failure Clinical Research Network. Ultrafiltration in decompensated heart failure with cardiorenal syndrome. N Engl J Med. 2012 Dec 13;367(24):2296-304. doi: 10.1056/NEJMoa1210357. Epub 2012 Nov 6. PMID 23131078
- [Derived] Rao VS, Ahmad T, Brisco-Bacik MA, Bonventre JV, Wilson FP, Siew ED, Felker GM, Anstrom KK, Mahoney DD, Bart BA, Tang WHW, Velazquez EJ, Testani JM. Renal Effects of Intensive Volume Removal in Heart Failure Patients With Preexisting Worsening Renal Function. Circ Heart Fail. 2019 Jun;12(6):e005552. doi: 10.1161/CIRCHEARTFAILURE.118.005552. Epub 2019 Jun 5. PMID 31163974
- [Derived] Kitai T, Grodin JL, Kim YH, Tang WH. Impact of Ultrafiltration on Serum Sodium Homeostasis and its Clinical Implication in Patients With Acute Heart Failure, Congestion, and Worsening Renal Function. Circ Heart Fail. 2017 Feb;10(2):e003603. doi: 10.1161/CIRCHEARTFAILURE.116.003603. PMID 28130379
- [Derived] de Denus S, Rouleau JL, Mann DL, Huggins GS, Cappola TP, Shah SH, Keleti J, Zada YF, Provost S, Bardhadi A, Phillips MS, Normand V, Mongrain I, Dube MP. A pharmacogenetic investigation of intravenous furosemide in decompensated heart failure: a meta-analysis of three clinical trials. Pharmacogenomics J. 2017 Mar;17(2):192-200. doi: 10.1038/tpj.2016.4. Epub 2016 Mar 1. PMID 26927285
- [Derived] Lala A, McNulty SE, Mentz RJ, Dunlay SM, Vader JM, AbouEzzeddine OF, DeVore AD, Khazanie P, Redfield MM, Goldsmith SR, Bart BA, Anstrom KJ, Felker GM, Hernandez AF, Stevenson LW. Relief and Recurrence of Congestion During and After Hospitalization for Acute Heart Failure: Insights From Diuretic Optimization Strategy Evaluation in Acute Decompensated Heart Failure (DOSE-AHF) and Cardiorenal Rescue Study in Acute Decompensated Heart Failure (CARESS-HF). Circ Heart Fail. 2015 Jul;8(4):741-8. doi: 10.1161/CIRCHEARTFAILURE.114.001957. Epub 2015 Jun 3. PMID 26041600
- [Derived] Mentz RJ, Stevens SR, DeVore AD, Lala A, Vader JM, AbouEzzeddine OF, Khazanie P, Redfield MM, Stevenson LW, O'Connor CM, Goldsmith SR, Bart BA, Anstrom KJ, Hernandez AF, Braunwald E, Felker GM. Decongestion strategies and renin-angiotensin-aldosterone system activation in acute heart failure. JACC Heart Fail. 2015 Feb;3(2):97-107. doi: 10.1016/j.jchf.2014.09.003. Epub 2014 Oct 31. PMID 25543972

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrafiltration: Participants will receive ultrafiltration
Period: Overall Study
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Started | 94 | 94
Completed | 73 | 72
Not Completed | 21 | 22

BASELINE CHARACTERISTICS:
Groups:
- Stepped Pharmacologic Care: Participants will receive stepped pharmacologic care
- Total: Total of all reporting groups
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration | Total
Number analyzed (Participants) | 94 | 94 | 188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 35 | 77
  >=65 years | 52 | 59 | 111
Age Continuous [Mean (Standard Deviation); unit: years] | 67.1 (13.7) | 68.9 (12.0) | 68.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 21 | 47
  Male | 68 | 73 | 141

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Creatinine
Time Frame: Change from Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 94 | 92
mg/dL | -0.04 (0.53) | 0.23 (0.70)

2. Secondary Outcome: Change in Glomerular Filtration Rate
Time Frame: Change from Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 94 | 92
mL/min | 1.67 (10.94) | 0.93 (14.60)

3. Secondary Outcome: Change in Serum Creatinine
Time Frame: Change from Baseline to Day 7
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 94 | 92
mg/dL | -0.00 (0.60) | 0.11 (0.89)

4. Secondary Outcome: Change in Glomerular Filtration Rate
Time Frame: Change from Baseline to Day 7
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 94 | 92
mL/min | 2.06 (9.32) | 1.82 (13.84)

5. Secondary Outcome: Changes in Weight
Time Frame: Change from Baseline to Day 1
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 90 | 88
lbs | -3.4 (5.2) | -4.4 (4.5)

6. Secondary Outcome: Changes in Weight
Time Frame: Change from Baseline to Day 2
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 94 | 91
lbs | -7.4 (8.6) | -8.8 (7.4)

7. Secondary Outcome: Change in Weight
Time Frame: Change from Baseline to Day 3
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 88 | 86
lbs | -10.8 (10.5) | -11.7 (7.7)

8. Secondary Outcome: Changes in Weight
Time Frame: Change from Baseline to Day 5
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 62 | 69
lbs | -15.6 (12.0) | -14.3 (10.0)

9. Secondary Outcome: Change in Weight
Time Frame: Change from Baseline to Day 6
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 51 | 59
lbs | -16.5 (15.3) | -15.7 (11.8)

10. Secondary Outcome: Cumulative Net Fluid Loss
Time Frame: Randomization through Day 1
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 94 | 93
mL | 1714.1 (1400.2) | 2193.6 (1554.9)

11. Secondary Outcome: Cumulative Net Fluid Loss
Time Frame: Randomization through Day 2
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 92 | 93
mL | 3814.2 (2384.2) | 4705.8 (2626.9)

12. Primary Outcome: Change in Weight
Time Frame: Change from Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 94 | 93
lbs | -12.1 (11.3) | -12.6 (8.5)

13. Secondary Outcome: Cumulative Net Fluid Loss
Time Frame: Randomization through Day 3
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 89 | 90
mL | 5706.8 (3490.6) | 6257.1 (3519.7)

14. Secondary Outcome: Cumulative Net Fluid Loss
Time Frame: Randomization through Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 79 | 81
mL | 7081.5 (4183.4) | 7443.0 (4328.7)

15. Secondary Outcome: Cumulative Net Fluid Loss
Time Frame: Randomization through Day 5
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 63 | 69
mL | 8358.8 (5034.5) | 8308.4 (5178.1)

16. Secondary Outcome: Cumulative Net Fluid Loss
Time Frame: Randomization through Day 6
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 53 | 55
mL | 9700.7 (6945.9) | 9822.1 (6001.7)

17. Secondary Outcome: Cumulative Net Fluid Loss
Time Frame: Randomization through Day 7
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 40 | 47
mL | 11659.6 (9142.0) | 10595.1 (7097.4)

18. Secondary Outcome: Dyspnea Visual Analog Scale
Description: Scale range: -100 , +100
  -100=worse, +100=better
Time Frame: Change from Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 88 | 83
units on a scale | 20.5 (27.8) | 16.5 (29.2)

19. Secondary Outcome: Change in Global Visual Analog Scale
Description: Scale range: -100 , +100
  -100=worse, +100=better Participants asked to mark their global well being on a 10 cm vertical line, with the top labeled "best you have ever felt" and the bottom labeled "worst you have ever felt".
Time Frame: Change from Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 87 | 81
units on a scale | 22.8 (25.8) | 13.7 (27.9)

20. Secondary Outcome: Change in Dyspnea Visual Analog Scale
Description: Scale range: -100 , +100
  -100=worse, +100=better
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 88 | 86
units on a scale | 22.8 (27.6) | 19.4 (31.4)

21. Secondary Outcome: Change in Global Visual Analog Scale
Description: as for outcome 19
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 87 | 86
units on a scale | 25.8 (30.2) | 16.9 (29.0)

22. Secondary Outcome: Change in Furosemide-Equivalent Dose
Description: Furosemide-Equivalent Dose is the dose bumetanide or torsemide converted to furosemide equivalent (Torsemide dose x 2,Bumetanide dose x 40)
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 92 | 89
mg | 2.2 (166.5) | -20.6 (116.0)

23. Secondary Outcome: Change in Blood Sodium Level
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 94 | 92
mEq/L | 0.00 (3.60) | -2.3 (3.51)

24. Secondary Outcome: Change in Blood Potassium Level
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 94 | 92
mEq/L | -0.23 (0.63) | 0.26 (0.70)

25. Secondary Outcome: Change in Blood Urea Nitrogen/Urea
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 94 | 93
mg/dL | 5.68 (18.29) | 12.54 (24.81)

26. Secondary Outcome: Change in Blood Bicarbonate Level
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 89 | 84
mEq/L | 3.29 (3.82) | -1.01 (4.17)

27. Secondary Outcome: Change in Blood Hemoglobin Level
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 89 | 93
g/dL | 0.38 (0.76) | -0.01 (0.92)

28. Secondary Outcome: Change in Blood Sodium Level
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 94 | 92
mEq/L | -0.49 (3.70) | -2.02 (4.11)

29. Secondary Outcome: Change in Blood Potassium Level
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 94 | 92
mEq/L | -0.14 (0.60) | 0.27 (0.75)

30. Secondary Outcome: Change in Blood Urea Nitrogen/Urea
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 94 | 93
mg/dL | 7.23 (20.69) | 13.81 (23.91)

31. Secondary Outcome: Change in Blood Bicarbonate Level
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 89 | 84
mEq/L | 3.07 (4.50) | -0.70 (5.03)

32. Secondary Outcome: Change in Blood Hemoglobin Level
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 89 | 93
g/dL | 0.35 (0.94) | -0.02 (0.96)

33. Secondary Outcome: Change in Blood Cystatin C
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 85 | 81
mg/L | 0.14 (0.52) | 0.22 (0.52)

34. Secondary Outcome: Change in Uric Acid
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 85 | 80
mg/dL | 1.06 (1.44) | -0.23 (1.67)

35. Secondary Outcome: Change in Blood N- Terminal Pro- BNP
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 84 | 79
pg/mL | -978.61 (2902.06) | -814.45 (9238.91)

36. Secondary Outcome: Change in Plasma Renin Activity
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ng/mL/hr
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 85 | 81
ng/mL/hr | 5.78 (45.65) | 12.67 (31.32)

37. Secondary Outcome: Change in Blood High Sensitivity Troponin I
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 84 | 81
pg/mL | 47.38 (369.85) | -38.95 (1027.37)

38. Secondary Outcome: Change in Blood Aldosterone
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 86 | 81
pg/mL | -109.13 (489.50) | -3.07 (485.40)

39. Secondary Outcome: Change in Blood Procollagen III N-terminal Propepide
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 86 | 81
ug/L | 0.22 (4.69) | -0.64 (4.02)

40. Secondary Outcome: Change in Blood Endothelin-1
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 83 | 78
pg/mL | -0.76 (1.70) | -1.13 (3.20)

41. Secondary Outcome: Change in Blood High Sensitivity C-Reactive Protein
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 85 | 81
mg/L | -1.71 (46.14) | 1.89 (28.60)

42. Secondary Outcome: Change in Blood Carboxy-terminal Telopeptide of Collagen Type I
Time Frame: Baseline to Day 4
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 83 | 76
ug/L | 7.63 (11.93) | 9.07 (13.46)

43. Secondary Outcome: Change in Blood Cystatin C
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 86 | 83
mg/L | 0.12 (0.48) | 0.09 (0.66)

44. Secondary Outcome: Change in Blood Uric Acid
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 86 | 82
mg/dL | 1.10 (1.85) | -0.15 (2.07)

45. Secondary Outcome: Change in Blood N Terminal Pro-Natriuretic Peptide
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 86 | 83
pg/mL | -1071.88 (3309.45) | -740.82 (8604.86)

46. Secondary Outcome: Change in Plasma Renin Activity
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ng/mL/hr
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 86 | 83
ng/mL/hr | 2.58 (40.70) | 11.40 (32.75)

47. Secondary Outcome: Change in Blood High Sensitivity Troponin I
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 86 | 83
pg/mL | 37.28 (350.45) | -37.16 (1231.12)

48. Secondary Outcome: Change in Blood Aldosterone
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 87 | 83
pg/mL | -74.26 (507.96) | 68.13 (624.35)

49. Secondary Outcome: Change in Blood Procollagen III N-terminal Propepide
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 87 | 83
ug/L | -0.07 (5.90) | -0.93 (3.54)

50. Secondary Outcome: Change in Blood Endothelin-1
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 85 | 83
pg/mL | -0.69 (1.85) | -1.24 (3.22)

51. Secondary Outcome: Change in Blood Carboxy-terminal Telopeptide of Collagen Type I
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 85 | 83
ug/L | 10.21 (15.79) | 10.54 (15.04)

52. Secondary Outcome: Change in Blood High Sensitivity C-Reactive Protein
Time Frame: Baseline to Day 7/Discharge
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 86 | 83
mg/L | -6.39 (48.56) | 2.18 (37.72)

53. Secondary Outcome: Weight Change
Time Frame: Baseline to Day 30
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 73 | 68
lbs | -15.9 (22.4) | -13.4 (21.0)

54. Secondary Outcome: Change in Furosemide-Equivalent Dose
Description: as for outcome 22
Time Frame: Baseline to Day 30
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 78 | 74
mg | 9.8 (188.3) | 27.3 (120.1)

55. Secondary Outcome: Creatinine Change
Time Frame: Baseline to Day 30
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 75 | 70
mg/dL | -0.25 (0.68) | -0.12 (0.59)

56. Secondary Outcome: Glomerular Filtration Rate Change
Time Frame: Baseline to Day 30
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 75 | 70
mL/min | 7.95 (11.85) | 6.07 (16.13)

57. Secondary Outcome: Weight Change
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 66 | 63
lbs | -17.2 (21.1) | -15.4 (23.1)

58. Secondary Outcome: Change in Furosemide-Equivalent Dose
Description: as for outcome 22
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 73 | 72
mg | -12.4 (122.5) | 8.8 (128.5)

59. Secondary Outcome: Best Available Serum Creatinine Change
Description: Core laboratory when available. If not available, local laboratory results were used.
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 67 | 70
mg/dL | -0.28 (0.61) | -0.12 (0.67)

60. Secondary Outcome: Best Available Glomerular Filtration Rate Change
Description: Core laboratory when available. If not available, local laboratory results were used.
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 67 | 70
mL/min | 8.86 (13.26) | 5.63 (16.49)

61. Secondary Outcome: Change in Blood Uric Acid
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 56 | 54
mg/dL | -0.31 (2.28) | -0.54 (2.60)

62. Secondary Outcome: Change in Blood Cystatin C
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 56 | 55
mg/L | -0.18 (0.48) | -0.03 (0.60)

63. Secondary Outcome: Change in Blood N Terminal Pro - B Natriuretic Peptides
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 56 | 55
pg/mL | -490.56 (5638.86) | -937.69 (7389.14)

64. Secondary Outcome: Change in Plasma Renin Activity
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ng/mL/hr
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 56 | 55
ng/mL/hr | -2.18 (41.12) | 0.54 (20.48)

65. Secondary Outcome: Change in Blood High Sensitivity Troponin I
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 56 | 55
pg/mL | -17.48 (106.70) | -73.58 (511.98)

66. Secondary Outcome: Change in Blood Aldosterone
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 57 | 55
pg/mL | -6.91 (672.21) | 40.35 (471.50)

67. Secondary Outcome: Change in Blood Procollagen III N-terminal Propepide
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 57 | 56
ug/L | 0.75 (5.25) | 0.58 (6.02)

68. Secondary Outcome: Change in Blood Endothelin-1
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 56 | 55
pg/mL | -0.82 (1.58) | -1.32 (3.98)

69. Secondary Outcome: Change in Blood High Sensitivity C-Reactive Protein
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 56 | 55
mg/L | -13.62 (59.58) | 1.99 (44.92)

70. Secondary Outcome: Change in Blood Carboxy-terminal Telopeptide of Collagen Type I
Time Frame: Baseline to Day 60
Population: Participants analyzed consisted of those participants who had the endpoint data available to be derived.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Number analyzed (Participants) | 56 | 55
ug/L | 2.24 (13.44) | 4.57 (27.84)

ADVERSE EVENTS:
Arm/Group | Stepped Pharmacologic Care | Ultrafiltration
Serious Adverse Events (participants affected / at risk) | 54/94 | 68/94
Other Adverse Events (participants affected / at risk) | 0/94 | 0/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stepped Pharmacologic Care (N=94) | Ultrafiltration (N=94)
Anaemia (Blood and lymphatic system disorders) | 5 | 6
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 2
Cardiac Failure (Cardiac disorders) | 17 | 16
Cardiac Failure Acute (Cardiac disorders) | 12 | 15
Cardiac Failure Chronic (Cardiac disorders) | 0 | 2
Pulseless Electrical Activity (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Ventricular Fibrillation (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 2
Renal Failure (Renal and urinary disorders) | 11 | 10
Renal Failure Acute (Renal and urinary disorders) | 3 | 6
Renal Failure Chronic (Renal and urinary disorders) | 2 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 1
Renal Tubular Necrosis (Renal and urinary disorders) | 0 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No